CLINICAL TRIAL: NCT03617913
Title: Phase II Study Evaluating Combination Chemotherapy + Radiotherapy (RT) With Avelumab in Muscle Invasive Bladder Cancer
Brief Title: Avelumab in Combination With Fluorouracil and Mitomycin or Cisplatin and Radiation Therapy in Treating Participants With Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1752; NCI-2018-01539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1752 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2018-07-26; First posted 2018-08-07 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2021-03

CONDITIONS: Bladder Carcinoma Infiltrating the Muscle of the Bladder Wall; Stage II Bladder Cancer AJCC v8; Stage II Renal Pelvis Cancer AJCC v8; Stage II Ureter Cancer AJCC v8; Stage II Urethral Cancer AJCC v8; Stage III Bladder Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8; Urethral Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — avelumab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Mitomycin; Mitozytrex; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (avelumab, chemotherapy, radiation therapy) (Experimental): Participants receive avelumab IV over 60 minutes every 14 days for a total of 10 courses in the absence of disease progression or unacceptable toxicity. Beginning 29 days after the first dose of avelumab, participants receive either fluorouracil IV on days 1-5 and 16-20 during RT and mitomycin IV on day 1 of course 3, or cisplatin IV starting on day 1 of courses 3-5 for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Cisplatin; Drug: Fluorouracil; Drug: Mitomycin; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Mitomycin — Given IV
  Other Names: Ametycine; MITO; MITO-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies the side effects of avelumab and how well it works in combination with fluorouracil and mitomycin or cisplatin and radiation therapy in treating participants with muscle-invasive bladder cancer. Monoclonal antibodies, such as avelumab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as fluorouracil, mitomycin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Giving avelumab with chemotherapy and radiotherapy may work better in treating participants with muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete response rate of concurrent chemotherapy radiation treatment combined with avelumab for patients with muscle invasive bladder cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity (adverse event profile) of concurrent chemotherapy radiation treatment combined with avelumab.

II. To evaluate quality of life (QoL) at 1 year of concurrent chemotherapy radiation treatment combined with avelumab.

III. To evaluate progression-free survival and relapse-free survival at 1 year with concurrent chemotherapy radiation treatment combined with avelumab.

CORRELATIVE OBJECTIVES:

I. To explore biomarkers that may predict response to avelumab in the muscle invasive population.

II. To evaluate the association of tumor mutational burden with response to concurrent chemo- radiation and immunotherapy.

III. To evaluate whether concurrent chemoradiation and immunotherapy after maximal transurethral resection of bladder tumor (TURBT) is associated with a decrease in circulating Bim+CD11a^high PD-1+CD8+ T-cells and myeloid-derived suppressor cells (MDSCs).

OUTLINE:

Participants receive avelumab intravenously (IV) over 60 minutes every 14 days for a total of 10 courses in the absence of disease progression or unacceptable toxicity. Beginning 29 days after the first dose of avelumab, participants receive either fluorouracil IV on days 1-5 and 16-20 during radiation therapy (RT) and mitomycin IV on day 1 of course 3, or cisplatin IV starting on day 1 of courses 3-5 for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of T2-T4a N0M0 (American Joint Committee on Cancer [AJCC] 8th edition) with predominant urothelial carcinoma. Mixed histologies are acceptable provided urothelial carcinoma is the predominant histology. Small cell urothelial carcinoma is excluded.
* Cystoscopy with maximal TURBT performed =< 70 days of study registration. NOTE: Both completely resectable or partially resectable tumors are eligible as long as the treating urologist attempted complete resection. Exam under anesthesia needs to be performed and documented.
* Absolute neutrophil count (ANC) >= 1500/mm^3 =< 28 days prior to registration.
* Platelets (PLT) 100,000/mm^3 =< 28 days prior to registration.
* Total bilirubin =< 1.5 upper limit of normal (ULN) =< 28 days prior to registration.
* Aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement) =< 28 days prior to registration.
* Alanine aminotransferase (ALT) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement) =< 28 days prior to registration.
* Hemoglobin (Hgb) >= 9 gm/dl =< 28 days prior to registration.
* Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula =< 28 days prior to registration.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS 0, 1, 2).
* Ability to provide informed written consent.
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study).
* Life expectancy >= 6 months.
* Negative serum pregnancy test done =< 14 days prior to registration, for women of childbearing potential only.

Exclusion Criteria:

* Patients with locally advanced unresectable (T4b) or metastatic urothelial carcinoma (N1M0-1) as assessed on baseline radiographic imaging obtained =< 70 days prior to study registration. The required radiographic imaging includes:

  * Abdomen/pelvis computed tomography (CT) or magnetic resonance imaging (MRI) scan
  * Chest x-ray or CT scan.
* Patients with concurrent urothelial carcinoma and/or related variants anywhere outside bladder

  * NOTE: Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
* A prior or concurrent malignancy of any other site or histology unless the patient has been disease-free for > 2 years prior to registration except for:

  * Non-melanoma skin cancer and/or localized prostate cancer (T2 a or b , Gleason < 3+4) or carcinoma in situ of the uterine cervix which has been adequately treated =< 2 years prior to registration
  * Or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai stage 0, prostate cancer with Gleason score =< 3+4, and prostate-specific antigen [PSA] =< 10 mg/mL, etc.).
* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies =< 4 weeks prior to registration, or who have not recovered from the side effects of such therapy.

  * EXCEPTION: Except single dose intravesical chemotherapy administered after TURBT.
* Patients who have received prior therapy with immune checkpoint inhibitors (e.g. anti-PD-1, anti-PD-L1, anti-LAG3, anti-CTLA-4, anti-TIM3) or immune co-stimulatory molecules (e.g. anti-CD137, anti-OX40, anti-GITR) directed agents.
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury =< 4 weeks prior to registration, or who have not recovered from side effects of such procedure or injury prior to registration.

  * NOTE: Patients who have had minor procedures (i.e. TURBT) or percutaneous biopsies prior to registration are eligible.
* Patients with history of cirrhosis, alcoholic or non-alcoholic steatohepatitis (NASH), auto-immune hepatitis, or previous grade 3-4 drug-related hepatitis.
* Patient with history of prior solid organ or allogeneic bone marrow transplant.
* Clinically significant cardiac diseases, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias.
  * Clinically significant resting bradycardia.
  * Any of the following =< 3 months prior to registration: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), congestive heart failure (CHF), cerebrovascular accident (CVA), transient ischemic attack (TIA), pulmonary embolism (PE).
  * Uncontrolled hypertension defined by a systolic blood pressure (SBP) >= 160 mm Hg and/or diastolic blood pressure (DBP) >= 100 mm Hg, with or without anti-hypertensive medication(s).
* History of untreated human immunodeficiency virus (HIV)

  * NOTE: There is no requirement to screen patients for HIV. Patients with history of HIV infection are allowed if on effective highly active antiretroviral therapy (HAART) therapy and CD4 count more than 250.
* History of active hepatitis B infection

  * NOTE: There is no requirement to screen patients for hepatitis B.
* Known diagnosis of any condition (i.e. post-hematopoietic or organ transplant, rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy.

  * NOTE: Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted. For questions, please consult the study chair.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Pregnant or breast-feeding women.
* Women of child-bearing potential, who are biologically able to conceive, and not employing two forms of highly effective contraception. Highly effective contraception must be used throughout the trial and up to 8 weeks after the last dose of study drug (e.g. male condom with spermicidal; diaphragm with spermicide; intra-uterine device). Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 14 days prior to registration.
* Fertile males not willing to use contraception, as stated above.
* Patients unwilling or unable to comply with the protocol.
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0 grade >= 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parminder Singh, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Avelumab and Cisplatin IV: Participants received avelumab IV over 60 minutes every 14 days for a total of 10 courses in the absence of disease progression or unacceptable toxicity. Beginning 29 days after the first dose of avelumab, participants received 35 mg/m^2/day cisplatin IV starting on day 1 of courses 3-5 for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Avelumab and Cisplatin IV
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants registered were included in this analysis.
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 65 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Complete Response (At 6 Months)
Description: Patients enrolled will have non-measurable disease based on imaging at baseline. Patients will be assessed for a response after 6 months of treatment using the results of a biopsy and cytology test. A complete response (CR) is defined as having a negative biopsy and negative urine cytology at 6 months from registration after finishing of concurrent RT and immunotherapy. Imaging of abdomen and pelvis confirming no systemic disease within 4 weeks of cystoscopy will be completed.
  The proportion of patients reporting a CR is reported here with confidence intervals for the true success proportion using the binomial distribution.
Time Frame: At 6 months from registration
Population: All patients who registered and began protocol treatment are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 2
proportion of participants | 0.5 [0.013 to 0.987]

2. Secondary Outcome: Adverse Events Per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. The number of patients reporting a grade 3+ adverse event regardless of attribution is reported here.
Time Frame: Up to 12 months
Population: All patients who were registered, received protocol treatment, and were assessed for adverse events were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 2
Participants
  Grade 3+ Adverse Event | 2
  Grade 4+ Adverse Event | 0

3. Secondary Outcome: Patient-reported Outcomes (European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-30
Description: EORTC QLQ-C30 is a 30-item patient-reported questionnaire. 28 of the 30 items are measured on a 1-4 scale (1=not at all; 4=very much) with the remaining two items (overall health and overall quality of life) scored on a 1-7 numeric analogue scale (1=very poor; 7=excellent). The recall period for the EORTC QLQ-C30 is one week.
  Changes from baseline will be statistically tested using paired t-tests, and standardized response means (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's (2002) adjustment) using Cohen's (1988) cut-offs: <0.20 = trivial; 0.20-<0.50 = small; 0.50-<0.80 = moderate; and >=/0.80 = large. Correlation between outcomes will employ Pearson and/or Spearman correlations at individual time points.
Time Frame: Baseline to 12 months
Population: All patients who were registered, treated, and completed the EORTC QLQ assessment at baseline and post-therapy were included in this analysis
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient-reported Outcomes (European Organization for Research and Treatment of Cancer [EORTC] EORTCQOL-Muscle-Invasive Bladder Cancer Module [BLM]30
Description: EORTC QLQ-BLM30 is a 30-item questionnaire for patients with muscle invasive bladder cancer (T2, T3, T4a and T4b). The muscle-invasive bladder cancer module contains additional items assessing urostomy problems, problems associated with the use of a catheter, and body image.
  Changes from baseline will be statistically tested using paired t-tests, and standardized response means (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's (2002) adjustment) using Cohen's (1988) cut-offs: <0.20 = trivial; 0.20-<0.50 = small; 0.50-<0.80 = moderate; and >=/0.80 = large. Correlation between outcomes will employ Pearson and/or Spearman correlations at individual time points.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the time of progression or death. This study will not use RECIST criteria to evaluate response or progression. The patients enrolled will have non-measurable disease on imaging and response will be evaluated with biopsy or cytology. Progression is defined as progression in T stage, N stage or M stage both clinically or radiologically. Histological confirmation of metastatic disease is at the discretion of the treating provider. The median time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to time of first documentation of progression or death from any cause, assessed up to 12 months
Population: All patients who registered and were treated are included in this analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 2
years | NA [NA to NA] — Too few events have occurred to obtain a median or a 95% CI.

6. Secondary Outcome: Recurrence-free Survival
Description: Recurrence-free survival is defined as the time from registration to the time of recurrence or death. Recurrence is defined as having histologically proven first appearance of muscle invasive bladder cancer, clinical evidence of metastatic disease, or treatment with radical cystectomy or radiation to the bladder, or death due to any cause after they were confirmed remission at 6 month evaluation.
  The median time will be estimated using the method of Kaplan-Meier.
Time Frame: From documented complete response to the first documentation of recurrence, assessed up to 12 months
Population: All patients who were registered, treated, and were assessed as having a Complete Response (CR) are eligible for this analysis. This endpoint can only be analyzed if more than one patient is eligible.
Arm/Group | Avelumab and Cisplatin IV
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Relationship of PD-L1 (SP263 and SP142), CD8+ by Immunohistochemistry
Description: Association of Bim (BCL-2-interacting mediator of cell death) expression will be evaluated at using the baseline tissue specimen and explored in relation to 6 months post-registration response and subsequently in relation to other clinical outcomes such as tumor response and adverse event incidence using two-way tables and analyzed using Fisher's exact tests.
Time Frame: Up to 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Tumor Mutational Burden With Response to Concurrent Chemo- Radiation and Immunotherapy
Description: Association of Bim expression will be evaluated at using the baseline tissue specimen and explored in relation to 6 months post-registration response and subsequently in relation to other clinical outcomes such as tumor response and adverse event incidence using two-way tables and analyzed using Fisher's exact tests. Expression of immune signatures by RNA-seq expression (using the baseline tissue specimen) will be evaluated at baseline and explored in relation to clinical outcomes such as progression-free survival, tumor response, and adverse event incidence using two-way tables and box plots and analyzed using Fisher's exact tests or logistic regression methods, as appropriate.
Time Frame: Up to 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Evaluate Whether Concurrent Chemoradiation and Immunotherapy After Maximal TURBT is Associated With a Decrease in Circulating Bim+CD11ahighPD-1+CD8+ T-cells and MDSCs.
Description: as for outcome 8
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed at the end of every 14 day cycle during treatment, up to 12 cycles.
Description: Adverse Events were assessed at the end of every 14 day cycle during treatment, up to 12 cycles.
Arm/Group | Avelumab and Cisplatin IV
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab and Cisplatin IV (N=2)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab and Cisplatin IV (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (14)
Diarrhea (Gastrointestinal disorders) | 1 (9)
Nausea (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (13)
Pain (General disorders) | 1 (7)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 2 (25)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03617913/Prot_SAP_000.pdf